CLINICAL TRIAL: NCT05617430
Title: An Exploratory Study to Evaluate the Efficacy and Safety of Hepatic Arterial Infusion Chemotherapy (HAIC) Combine With Sintilimab and Bevacizumab for BCLC-C Hepatocellular Carcinoma
Brief Title: Combination Therapy of HAIC, Sintilimab and Bevacizumab for Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT22623
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Folfox protocol; Therapeutics; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC + Sintilimab + Bevacizumab (Experimental): HAIC combine with Sintilimab and bevacizumab biosimilar
  Interventions: Drug: HAIC; Drug: Sintilimab; Drug: Bevacizumab Biosimilar IBI305

INTERVENTIONS:
Drug: HAIC — Oxaliplatin: 85mg/m2 , Day 1 Leucovorin: 200mg/m2, Day 1 Fluorouracil: 400mg/m2, Day1 and 2400mg/m2 continuous arterial perfusion for 46h.
  Q3W
  Other Names: hepatic arterial infusion (HAI) of oxaliplatin, fluorouracil, leucovorin (FOLFOX) treatment (Q3W)
Drug: Sintilimab — 200mg IV d1, Q3W
  Other Names: IBI308
Drug: Bevacizumab Biosimilar IBI305 — 7.5mg/kg IV d1, Q3W
  Other Names: IBI305

SUMMARY:
This is a single-arm, exploratory study to evaluate the efficacy and safety of HAIC in combination with sintilimab and bevacizumab in the first line treatment of patients with BCLC-C hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent should be signed before implementing any trial-related procedures 2. ECOG PS scores 0-1 3. Histologically/cytologically confirmed HCC or cirrhosis meeting the clinical diagnostic criteria of HCC by American Association for the Study of Liver Diseases (AASLD) 4. Barcelona Clinic Liver Cancer (BCLC) stage C 5. Newly diagnosed HHC patients without any previous treatment for the tumor 6. Child Pugh score of ≤ 7. 7. Estimated survival > 12 weeks 8. At least one measurable lesion according to RECIST V1.1 9. Sufficient organ and bone marrow functions, with the laboratory test values within 7 days before the enrollment meeting the following requirements (no blood components, cell growth factors, albumin, and other drugs via intravenous or subcutaneous administrations are allowed for correction treatment within the first 14 days after the laboratory test results are obtained). The specific information is as follows:

1. Routine blood test: absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 75 × 109/L; hemoglobin (HGB) ≥ 9.0 g/dL.
2. Hepatic function: total bilirubin (TBIL) ≤ 3 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN; serum albumin ≥ 28 g/L; alkaline phosphatase (ALP) ≤ 5 × ULN.
3. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN or clearance of creatinine (CCr) ≥ 50 mL/min (Cockcroft Gault formula); urinalysis results showing urine protein < 2+; patients whose baseline urinalysis results show urine protein ≥ 2+ should undergo 24 h urine collection and the 24 h urine protein quantitation test result should be lower than 1 g.
4. Blood coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

10. Female patients of childbearing age or male patients with female sexual partners of childbearing age should take effective contraceptive measures throughout the treatment and 6 months after the last dose.

Exclusion Criteria:

1. Histologically/cytologically confirmed fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and cholangiocarcinoma.
2. History of hepatic encephalopathy or liver transplantation.
3. Symptomatic pleural effusion, ascites, and pericardial effusion that require drainage.
4. Acute or chronic active hepatitis B or C infection; hepatitis B virus (HBV) DNA > 2000 IU/mL or 104 copies/mL; hepatitis C virus (HCV) RNA > 103 copies/mL; hepatitis B surface antigen (HbsAg) and anti HCV antibody positive concurrently.
5. Presence of metastasis to the central nervous system.
6. Presence of bleeding events from esophageal or gastric varices caused by portal hypertension within the past 6 months. Presence of known severe (G3) varicose veins in endoscopy within 3 months before the first dose. Evidence of portal hypertension (including the finding of splenomegaly in imaging studies) with a high risk of bleeding assessed by the investigator.
7. Presence of any life-threatening bleeding events within the past 3 months, including the need for transfusion, surgery or local treatment, and continuous medication therapy.
8. Any arterial/venous thromboembolic events within 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient cerebral ischemic attack, pulmonary embolism, deep vein thrombosis, or any other history of serious thromboembolism. Presence of implantable venous port or catheter derived thrombosis, or superficial venous thrombosis, barring stable thrombosis following the conventional anticoagulation treatment. Prophylactic use of low dose low molecular weight heparin (e.g., enoxaparin 40 mg/day) is permitted.
9. Involvement of both the main portal vein and the left and right branches by portal vein tumor thrombus, or of both the main trunk and the superior mesenteric vein concurrently. Presence of tumor thrombus of inferior vena cava.
10. A 10-day consecutive dosing of aspirin (> 325 mg/day) or other drugs, e.g., dipyridamole and clopidogrel, known to inhibit the platelet function within 2 weeks before the first dose.
11. Uncontrolled hypertension (systolic greater than 140 mmHg or diastolic greater than 90 mmHg) after the optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
12. Toxicity (excluding alopecia, events not clinically significant, and asymptomatic laboratory abnormalities) caused by previous therapy that has not yet resolved to grade 0 or 1 (National Cancer Institute Common Terminology Criteria for Adverse Events V5.0 (NCI CTCAE V5.0)) before the first dose of study drugs.
13. Symptomatic congestive cardiac failure (NYHA Class II IV). Symptomatic or poorly controlled arrhythmia. History of congenital long QT syndrome or corrected QTc > 500 ms (calculated using Fridericia formula) during screening.
14. Serious hemorrhagic tendency or coagulopathy, or currently receiving thrombolytic therapy.
15. History of gastrointestinal perforation and/or fistula, history of bowel obstruction (including incomplete bowel obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection accompanied with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within the past 6 months.
16. Receipt of immunosuppressants within 4 weeks before the first dose, excluding local glucocorticoids administered by nasal, inhaled, or other topical routes, or systemic glucocorticoids of physiological doses (no more than 10 mg/day of prednisone or equivalents), while the temporary use of glucocorticoids for preventing allergies or treating dyspneic symptoms of such diseases as asthma and chronic obstructive pulmonary disease is permitted.
17. Receipt of a live attenuated vaccine within 4 weeks before the first dose or planned to receive a live attenuated vaccine during the study.
18. Receipt of major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks before the first dose or having unhealed wounds, ulcers, or fractures. Receipt of tissue biopsy or other minor surgeries within 7 days before the first dose, barring venipuncture and catheterization for intravenous infusion.
19. Receipt of local treatment for liver cancer within 4 weeks before the first dose.
20. Receipt of systemic treatment with traditional Chinese medicines with cancer indications or immunomodulators (including thymosin, interferon, and interleukin, barring local use for controlling pleural fluid or ascites) within 2 weeks before the first dose.
21. Uncontrolled/uncorrectable metabolic disorders, other non malignant organ diseases, systemic diseases, or cancer related secondary diseases with the potential to cause a relatively high medical risk and/or survival evaluation uncertainties unsuitable for subject enrollment as judged by the investigator; other circumstances unsuitable for subject enrollment as judged by the investigator.
22. Other malignancies diagnosed within 5 years before the first dose, excluding radically treated basal cell carcinoma of skin, squamous cell carcinoma of skin, and/or radically resected carcinoma in situ. If other malignancies were diagnosed over 5 years pre dose, the liver lesions should still be subjected to pathological or cytological diagnosis even if they meet the clinical diagnostic criteria for HCC by AASLD; individuals with confirmed HCC can be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) per RECIST v1.1 | From baseline to primary completion date, about 18 months
  Defined as a duration from the date of initial treatment to disease progression or death of any cause

SECONDARY OUTCOMES:
The treatment-related adverse events (TRAEs) | From baseline to primary completion date, about 18 months
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0
Overall response rate (ORR) per RECIST v1.1 and mRECIST | From baseline to primary completion date, about 18 months
  Defined as the incidence of complete response and, partial response
Disease control rate (DCR) per RECIST v1.1 and mRECIST | From baseline to primary completion date, about 18 months
  Defined as the incidence of complete response, partial response and stable disease
Duration of response (DoR) per RECIST v1.1 and mRECIST | From baseline to primary completion date, about 18 months
  Defined as a duration from date of initial treatment to disease progression or death in patients who achieve complete or partial response
Overall survival (OS) | From baseline to primary completion date, about 18 months
  Defined as a duration from the date of initial treatment to death of any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No